CLINICAL TRIAL: NCT06500806
Title: The Effect of a Long-Term Schroth Exercise Program on the Severity of Scoliosis and Quality of Life in Adolescents With Adolescent Idiopathic Scoliosis Wearing a Brace: A Randomized Controlled Clinical Trial
Brief Title: Impact of Long-Term Schroth Exercises on Scoliosis Severity and Quality of Life in Braced AIS Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Hellenic University (Other)
Responsible Party: Principal Investigator, Dimitrios Lytras, Dimitrios Lytras, Principal Investigator, Senior Lecturer of Physiotherapy, International Hellenic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC-09/2022
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: Adolescent idiopathic scoliosis; Schroth exercises; Conservative treatment; Physiotherapy
MeSH Terms: interventions — Braces

STUDY DESIGN:
Intervention Model Description: This randomized clinical trial will be under the supervision of the Department of Physiotherapy at the School of Health Sciences, International Hellenic University. Participants will be adolescents aged 10 to 17 years with mild to moderate scoliosis (Cobb angle from 10° to 45°) who will be prescribed a brace. The participants will be randomly assigned to two groups. The intervention group will follow a supervised Schroth exercise program alongside brace use for 12 months, with sessions three times a week. The control group will receive only brace treatment and recommendations for physical activity. The intervention will last one year, with a follow-up six months after the end of the intervention (18th month)
Who Masked: Outcomes Assessor
Masking Description: A masked assessor will conduct the measurements
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scroth and brace Group (Experimental): Participants allocated to this group will receive bracing and Schroth exercises for 12 months
  Interventions: Other: Scroth and brace
- Brace group (Active Comparator): Participants in this group will follow brace treatment.
  Interventions: Device: Brace

INTERVENTIONS:
Other: Scroth and brace — Participants in this group will wear a brace and follow a 12-month Schroth exercise program three times a week. Sessions will be supervised by a physiotherapist and last 60 minutes, using equipment like foam blocks, exercise balls, and rods. Exercise intensity will gradually increase based on progress. The individualized Schroth exercises will aim to correct spinal deformity and include elongation, rotational correction, stretches, strengthening, and breathing exercises. These exercises will help patients maintain proper posture in daily activities and will be adapted to each participant's abilities, with varying difficulty and positions.
  Arms: Scroth and brace Group
Device: Brace — Participants in this group will follow only the brace treatment
  Arms: Brace group

SUMMARY:
Adolescent Idiopathic Scoliosis (AIS) affects individuals aged 10 to 18, leading to spinal deformity and vertebral rotation. The Schroth exercise method, combined with brace usage, has shown promise in reducing the Cobb angle and preventing further deformity. This study aims to evaluate the impact of a 12-month supervised Schroth exercise program on scoliosis severity and quality of life in adolescents with AIS. Eighty adolescents, aged 10 to 17, were divided into two groups: one group received Schroth exercises along with bracing, while the control group used only a brace. Measurements included the Cobb angle, Angle Trunk Rotation (ATR), and quality of life using the SRS-22 questionnaire, assessed at the start, after 12 months, and 18 months. Analysis used Multivariate Analysis of Covariance (MANCOVA), with p < 0.05 as the significance level. We expect that the addition of Schroth exercises to a 12-month bracing program will significantly improve scoliosis severity and quality of life.

DETAILED DESCRIPTION:
Background: Adolescent Idiopathic Scoliosis (AIS) affects individuals aged 10 to 18 and is characterized by spinal deformity in the frontal plane, three-dimensional distortion of the spine, and vertebral rotation. Exercises based on the Schroth method, along with the use of a brace, have been shown to reduce the Cobb angle and may prevent further spinal deformity.

Objective: This clinical study aims to investigate the impact of a 12-month supervised Schroth exercise program on the severity of scoliosis and the quality of life in adolescents diagnosed with AIS.

Method: In this study, 80 adolescents aged 10 to 17 with AIS who are prescribed a brace are divided into two groups: an intervention group and a control group. The intervention group participates in a supervised Schroth exercise regimen three times weekly for a year, in addition to wearing a brace. The control group uses only the brace. Measurements include the Cobb angle of the main curve, the sum of the curves via Surgimap 2.3.2.1 software, the Angle Trunk Rotation (ATR) with a scoliometer, and quality of life assessed through the SRS-22 questionnaire. These assessments are conducted at the start, after one year (12th month), and six months post-intervention (18th month). The data are analyzed using Multivariate Analysis of Covariance (MANCOVA), with statistical significance set at p < 0.05.

Expected Results: Previous studies indicate that Schroth exercises can reduce the Cobb angle and ATR in adolescents with AIS and slow the progression of spinal deformity. However, few studies have investigated the effects of Schroth exercises for periods longer than six months. It is anticipated that incorporating Schroth exercises into a 12-month brace treatment program will significantly improve both the severity of scoliosis and the quality of life for the participants.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Adolescent Idiopathic Scoliosis (AIS)
* Aged 10 to 17 years, inclusive of both genders
* Cobb angle between 10° and 45°
* Risser grade between 0 and 3
* Prescribed a scoliosis brace
* Written consent from their legal guardian for participation
* Ability to attend Schroth exercise sessions for one year

Exclusion Criteria:

* Any contraindication for exercise
* Scheduled surgery for scoliosis treatment
* Diagnosed intellectual disabilities (e.g., intellectual disability, autism)
* Diagnosed neurological or rheumatic conditions

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2024-07-28 (Actual); Study Completion 2024-07-28 (Actual)

PRIMARY OUTCOMES:
Changes in Cobb ankle | Pre-treatment, months: 12, 18
  An independent orthopedic physician will measure the Cobb angle using Surgimap 2.3.2.1 software. For each assessment, participants will undergo a radiological examination with a full spinal X-ray taken from an anteroposterior view while standing. The study will evaluate the Cobb angle of the primary curvature (the largest curve) as well as the total sum of the Cobb angles of all identified curves.
Changes in maximum Ankle Trunk Rotation | Pre-treatment, months: 12, 18
  The ATR (Angle of Trunk Rotation) will be measured using a scoliometer. For the ATR measurement, each participant will stand with their feet together in an upright position and perform a forward bend (Adam's forward bend test) until their back is parallel to the ground. The scoliometer will then be placed vertically along the spine at the level where the rib hump appears. In this study, the maximum ATR (ATR maximum) will be recorded.
Changes in quality of life with SRS - 22 questionnaire | Pre-treatment, months: 12, 18
  Participants' quality of life will be evaluated using the Scoliosis Research Society 22 (SRS-22) questionnaire. The SRS-22 is the standard tool for assessing the quality of life in individuals with scoliosis, comprising 22 questions across five categories: functionality (5 questions), pain (5 questions), self-image (5 questions), mental health (5 questions), and treatment satisfaction (2 questions). Responses are rated on a Likert scale from 1 to 5. The overall score is determined by averaging the subcategory scores, ranging from 1 (lowest) to 5 (highest), with higher scores indicating better quality of life. This study will use the Greek version of the questionnaire. The total SRS-22 score will be used to measure the quality of life. The Greek version has been shown to have high reliability and validity compared to the 36-Item Short Form Survey (SF-36).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physiotherapy, Faculty of Health Sciences International Hellenic University, Thessaloniki, Sindos Thessaloníki, Greece

IPD SHARING:
Plan to Share IPD: No